CLINICAL TRIAL: NCT03252327
Title: Effects of the Interventions Using Multiple Sensory Integrations on Relieving Pain and Distress in Preterm Infants During Peripheral Venous Puncture Procedures
Brief Title: Effects of the Interventions Using Multiple Sensory Integrations on Preterm Infants' Stress-Related Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Hsiang-Ping Wu, Principal Investigator, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2-106-05-080
Record Dates: First submitted 2017-08-08; First posted 2017-08-17 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Preterm Infants; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- routine care (No Intervention): Preterm infants in the control condition will receive only usual neonatal intensive care units (NICU) care
- Multiple Sensory Integrations(1) (Experimental): The sensory integrations are provided through combining the use of sensory integrations ( olfactory, taste, auditory or tactile).
  Interventions: Other: Multiple Sensory Integrations
- Multiple Sensory Integrations(2) (Experimental): The sensory integrations are provided through combining the use of sensory integrations ( olfactory, taste, auditory or tactile).
  Interventions: Other: Multiple Sensory Integrations
- Multiple Sensory Integrations(3) (Experimental): The sensory integrations are provided through combining the use of sensory integrations ( olfactory, taste, auditory or tactile).
  Interventions: Other: Multiple Sensory Integrations

INTERVENTIONS:
Other: Multiple Sensory Integrations — breast milk odor, oral expressed breast milk, heartbeat sounds, nonnutritive sucking.
  Arms: Multiple Sensory Integrations(1); Multiple Sensory Integrations(2); Multiple Sensory Integrations(3)

SUMMARY:
Frequent pain and distress may affect infants' brain and neural development, and highlight the need for relieve pain interventions. Peripheral venous puncture procedures are an important source of preterm infants' pain and distress. Brain development is mainly created by infant sensory experience. It becomes important, therefore, to relieve preterm infants' pain and distress using multiple sensory integrations during peripheral venous puncture procedures.The proposed 2-year study has specific aim: to compare the effects of different combination of sensory integrations on preterm infants' pain and distress before, during, and after peripheral venous puncture procedures.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) 28-37 weeks
* Post-menstrual age (PMA) 29-38 weeks
* Postnatal age 3-28 days
* Sable condition (NTISSscore ≦ 22)
* Apgar scores≧7 at 5 minutes after birth

Exclusion Criteria:

* Neurologic impairment
* Congenital anomalies
* Surgery
* Severe growth restriction at birth
* Severe medical conditions requiring treatments

Ages: 3 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2017-08-26 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Preterm infants' pain | 20-30 minutes (during peripheral venous puncture procedures)
  Premature Infant Pain Profile-Revised (PIPP-R) for pain, A score <7 suggests no or little pain, 7-12 mild to moderate pain and scores >12 indicate moderate to severe pain.

SECONDARY OUTCOMES:
preterm infants' physiological parameters:heart rate | 20-30 minutes (during peripheral venous puncture procedures)
  Heart rate will be recorded from ECG leads. Heart rate in beats per minute (mean of physiological parameters)
Preterm infants' physiological parameters:respiration rate | 20-30 minutes (during peripheral venous puncture procedures)
  Respiration rate will be recorded from ECG leads. Respiration rate in breaths per minute. (mean of physiological parameters)
Preterm infants' physiological parameters: oxygen saturation | 20-30 minutes (during peripheral venous puncture procedures)
  Oxygen saturation will be recorded from ECG leads. Oxygen saturation in % (mean of physiological parameters)
preterm infants' behavioral responses | 20-30 minutes (during peripheral venous puncture procedures)
  The infant behavioral responses will be measured by using an infant behavioral coding scheme. Behavioral data during venous puncture procedures will be collected using a real-time colour video recorder. Frequency ratios for pain and distress behaviors, include: facial activity (e.g. brow bulge, eye squeeze, nasolabial furrow), body movement, cry, transition between sleep and wake states.
preterm infants' duration of fussing and cry | 20-30 minutes (during peripheral venous puncture procedures)
  Fussing and crying will be record from the recording pen in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan